CLINICAL TRIAL: NCT05920213
Title: HELP Trial: Efficacy of L-Ornithine L-Aspartate and Polyethylene Glycol in Cirrhotic Patients With Overt Hepatic Encephalopathy
Brief Title: Efficacy of L-Ornithine L-Aspartate and Polyethylene Glycol in Cirrhotic Patients With Overt Hepatic Encephalopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, ZA, Associate professor, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: JSMU/IRB/2022/673
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Hepatic Encephalopathy Stage 2; Hepatic Encephalopathy Stage 3; Hepatic Encephalopathy Stage 4
Keywords: Lactulose / therapeutic use; Liver Cirrhosis / drug therapy; Ornithine; Aspartic Acid / therapeutic use; Liver Cirrhosis / complications; Hepatic Encephalopathy / drug therapy*; Polyethylene Glycols / therapeutic use*; Gastrointestinal Agents / therapeutic use*
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis | interventions — Polyethylene Glycols; Lactulose; ornithylaspartate

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants' attendants will also be masked and will give consent for the study in case the participant is admitted to the Intensive care unit and is not mentally stable to give consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactulose AND LOLA (Experimental): Lactulose which is the standard of care treatment will be administered with the experimental drug L-ornithine L-aspartate (LOLA).
  Interventions: Drug: Lactulose oral solution; Drug: L-ornithine L-aspartate
- Lactulose and PEG (Experimental): Lactulose which is the standard of care treatment will be administered with the experimental drug polyethylene glycol (PEG).
  Interventions: Drug: Polyethylene Glycols; Drug: Lactulose oral solution
- Lactulose (Active Comparator): This group will receive Lactulose only which is the standard of care treatment.
  Interventions: Drug: Lactulose oral solution

INTERVENTIONS:
Drug: Polyethylene Glycols — 280g/ 24 hours for 5 days
  Arms: Lactulose and PEG
Drug: Lactulose oral solution — 60-120 ml per day for 5 days
Drug: L-ornithine L-aspartate — 30g/24 hours in 3 divided doses for 5 days
  Arms: Lactulose AND LOLA

SUMMARY:
The goal of this clinical trial is to compare the efficacy of L-ornithine L-aspartate and Polyethylene Glycol in Cirrhotic Patients with Overt Hepatic Encephalopathy.

Participants will be asked to fill out a few questions on proforma that will obtain demographic information as well as information relating to the patient's health. Treatments that they will receive after inclusion in the study, will be the standard treatment (Lactulose) along with additional medication as part of our research (LOLA or Polyethylene glycol).

DETAILED DESCRIPTION:
This is a randomized control trial with the following objectives

* what is the efficacy of add-on LOLA therapy in patients of overt HE (Grade II and above) against the standard-of-care arm
* what is the efficacy of adding on polyethylene glycol (PEG) in overt HE (Grade II and above) against the standard-of-care arm

Randomization will be done using card randomization. three different color-coded cards will be kept. Any card will be randomly picked for the patient fulfilling inclusion criteria and will be treated according to the allocated treatment arm mentioned on the card

Patients will be diagnosed on the basis of Modified West Haven Criteria. For diagnosis and prognosis, the following tools will be used:

* Modified West Haven criteria and Glasgow coma scale will be used to assess the mental state.
* CLIF-C ADs and CLIF SOFA score will be used as a prognostic score for predicting mortality in hospitalized patients.
* Overt HE patients will be graded using the Hepatic encephalopathy grading instrument (HEGI).
* Child-Pugh classification and MELD scoring will be used to assess the severity of chronic liver disease and cirrhosis.

Written informed consent will be obtained from the immediate attendant of the patient. All ethical considerations will be followed.

Our research has been approved by Jinnah Sindh Medical University, Karachi. For this approval, the investigators have made every effort to ensure the confidentiality of research data collected from all our participants in this survey. The information collected will be stored with the investigators only in the form of de-identified information and will be retained in a secure place under lock and key. Any results that will be generated will be presented on a collective basis, and will not contain the participant's name or any other personal details.

Data entry and analysis will be done using SPSS Software version 23. Study analysis will be done using the principle of intention to treat. Primary and secondary outcomes will be studied among intervention and standard-of-care groups at a Confidence Interval of 95%. The chi-square test will be used to find the association of independent variables like age, gender, and HE grades with interventional therapies. Independent t-test will be used to compare mean scores between groups.

ELIGIBILITY:
Inclusion Criteria:

* Admitted cirrhotic patients above 18 years of age,
* diagnosed on clinical/ultrasound findings with HE (grade 2 or above) with or without precipitating factors.

Exclusion Criteria:

* Patients with hepatocellular carcinoma
* severe septicemia,
* active upper gastrointestinal bleeding and in a state of shock
* presence of underlying chronic renal failure (serum creatinine >1.5 mg/dl)
* presence of hepatorenal syndrome
* neurodegenerative disease
* patients with a head injury and drug intoxication
* acute superimposed liver injury
* advanced cardiac or pulmonary derangements
* end-stage renal disease
* pregnant or breastfeeding mothers
* patients who are on sedatives, antidepressants, or benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Patient recovery among all groups through a change in mental state. | Change will be assessed at enrollment.
  Change of at least one grade in the mental state based on the modified West Haven criteria and hepatic encephalopathy grading scale. A decrease in the grade will be a better outcome.
Patient recovery among all groups through a change in mental state. | Change will be assessed at 24 hours post enrollment.
  A change of at least one grade in the mental state based on the modified West Haven criteria and hepatic encephalopathy grading scale. A decrease in the grade will be a better outcome.
Patient recovery among all groups through a change in mental state. | A change will be assessed at 48 hours post enrollment.
  A change of at least one grade in the mental state based on the modified West Haven criteria and hepatic encephalopathy grading scale. A decrease in the grade will be a better outcome.
Patient recovery among all groups through a change in mental state. | A change will be assessed at 72 hours post enrollment.
  A change of at least one grade in the mental state based on the modified West Haven criteria and hepatic encephalopathy grading scale. A decrease in the grade will be a better outcome.
Patient recovery among all groups through a change in mental state. | A change will be assessed at 96 hours post enrollment.
  A change of at least one grade in the mental state based on the modified West Haven criteria and hepatic encephalopathy grading scale. A decrease in the grade will be a better outcome.
Patient recovery among all groups through a change in mental state. | A change will be assessed at 120 hours post enrollment.
  A change of at least one grade in the mental state based on the modified West Haven criteria and hepatic encephalopathy grading scale. A decrease in the grade will be a better outcome.
Patient recovery among all groups through a change in mental state. | A change will be assessed at 144 hours post enrollment.
  A change of at least one grade in the mental state based on the modified West Haven criteria and hepatic encephalopathy grading scale. A decrease in the grade will be a better outcome.

SECONDARY OUTCOMES:
A change in Quality of Life will be assessed through SF-36 | Quality of life will be assessed at 28th day post enrollment.
  A change in the quality of life will be assessed using a validated Urdu translation of the Rand Short Form 36 item survey (SF-36 U). The lower the score the more disability. The higher the score the less disability
A change in Quality of Life will be assessed through SF-36 | Quality of life will be assessed at 84th day post enrollment.
  A change in the quality of life will be assessed using a validated Urdu translation of the Rand Short Form 36 item survey (SF-36 U).The lower the score the more disability. The higher the score the less disability
A change in mortality rate | it will be inquired at 7th day post enrollment.
  It will be observed through weekly calls and monthly visits.
A change in mortality rate | it will be inquired at 28th day post enrollment.
  It will be observed through weekly calls and monthly visits.
A change in mortality rate | it will be inquired at 84th day post enrollment.
  It will be observed through weekly calls and monthly visits.

CONTACTS AND LOCATIONS:
Locations (6):
- Pakistan (6):
  - Bolan Medical Complex Hospital, Quetta, Balochistan
  - Sheikh Khalifa bin Zayed, Quetta, Balochistan
  - Nishtar Medical Univeristy and Hospital, Multan, Punjab Province
  - Sheikh Zayed Medical College/Hospital, Rahim Yar Khan, Punjab Province
  - Medical ICU, Jinnah Postgraduate Medical Centre, Karachi, Sindh
  - CMC hospital, Larkana, Sindh

IPD SHARING:
Plan to Share IPD: No